CLINICAL TRIAL: NCT02495571
Title: Pilot Observational Study, Assessing PCEF of the Voluntary and Reflex Cough in Patients With ALS
Brief Title: Assessment of Voluntary and Reflex Cough in Patients With ALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Irene Battel, Speech and Language Pathologist, IRCCS San Camillo, Venezia, Italy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TRSLA
Record Dates: First submitted 2015-06-30; First posted 2015-07-13 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: ALS; Cough
Keywords: ALS and Dysphagia; ALS and cough; cough reflex test
MeSH Terms: conditions — Cough; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALS Patients (Experimental): Study Group: Evaluation of the cough reflex and the voluntary cough by spirometer and nebulizer
  Interventions: Other: Cough Assessment in ALS Patients
- Healthy Subjects (Other): Control group matched by aged and sex with the study group
  Interventions: Other: Cough Assessment in ALS Patients

INTERVENTIONS:
Other: Cough Assessment in ALS Patients — 1. Volitional Cough assessment by spirometer:
     a) Peak Cough Espiratory Flow (PCEF)
  2. Cough Reflex Test a) Peak Cough Espiratory Flow (PCEF)

SUMMARY:
This study aims to assess the presence and the intensity of voluntary and cough reflex in patients with amyotrophic lateral sclerosis (ALS), comparing the results with the healthy control group. The assessment of the cough is fundamental to verify the mechanism of airways protection which is particularly compromised in ALS patients.

Objective parameters of voluntary and reflex cough would be measured by the spirometer. The reflex of cough would be elicited by a solution of citric acid through an ultrasonic nebulizer.

DETAILED DESCRIPTION:
Protocol:

1. Volitional Cough assessment by spirometer (Pony FX- Cosmed): a) Forced vital capacity (FVC); b) Volume Tidal; c) Maximum Espiratory Pressure (MEP); d) Maximum Inspiratory Pressure (MIP); e) Peak of Cough Expiratory Flow.
2. Cough Reflex would be trigged by the inhalation of 0.4M of citric acid solution using the ultrasonic nebulizer (MO-03 Norditalia Elettromedicali) connected with the spirometer and the nebulizer via a bidirectional valve. It would be measured the Peak of Cough Expiratory Flow.

Participants:

It would be recruited 60 subjects at the IRCCS Ospedale San Camillo Venezia (Italy). All participants have to provide informed consent independently. The study group is composed by thirty participants with diagnosis of ALS and the severity score of Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS). The control group consist of thirty healthy subjects matched by aged and sex with the study group.

Statistical consideration:

The variables measured will be summarized by means and standard deviations or by proportions. Numeric variables MIP-MEP-FVC-Vt-PCEF will be analyzed using the Shapiro-Wilk test to verify the normality of distribution. Depending on the outcome, for the comparison between groups will be used or the t-test (parametric) or the test of Mann Whitney (non-parametric) for independent samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS
* Consensus

Exclusion Criteria:

* Smokers
* Oxygen Therapy
* Invasive Ventilation
* Allergy of citrus
* Asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
PCEF of RC in ALS | 6 weeks
  Peak of Cough Expiratory Flow during reflex cough in ALS patients
PCEF of VC in ALS | 6 weeks
  Peak of Cough Expiratory Flow during volitional cough in ALS patients
PCEF of RC in healthy subjects | 6 weeks
  Peak of Cough Expiratory Flow during reflex cough in healthy subjects
PCEF of VC in healthy subjects | 6 weeks
  Peak of Cough Expiratory Flow during during volitional cough in healthy subjects

SECONDARY OUTCOMES:
PCEF of VC in ALS and control group | 8 weeks
  Comparison of PCEF of the voluntary cough between the 2 groups

OTHER OUTCOMES:
PCEF of RF in ALS and control group | 8 weeks
  Comparison of PCEF of the reflex cough between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: IRENE BATTEL, Principal Investigator — IRCCS San Camillo, Venezia, Italy
Locations (1):
- Fondazione Ospedale San Camillo IRCCS, Venice, Venice, Italy

REFERENCES:
- [Background] Widdicombe JG, Addington WR, Fontana GA, Stephens RE. Voluntary and reflex cough and the expiration reflex; implications for aspiration after stroke. Pulm Pharmacol Ther. 2011 Jun;24(3):312-7. doi: 10.1016/j.pupt.2011.01.015. Epub 2011 Feb 19. PMID 21338708
- [Background] Luchesi KF, Kitamua S, Mourao LF. Amyotrophic Lateral Sclerosis survival analysis: Swallowing and non-oral feeding. NeuroRehabilitation. 2014;35(3):535-42. doi: 10.3233/NRE-141149. PMID 25238863
- [Background] Zoccolella S, Beghi E, Palagano G, Fraddosio A, Samarelli V, Lamberti P, Lepore V, Serlenga L, Logroscino G; SLAP registry. Predictors of delay in the diagnosis and clinical trial entry of amyotrophic lateral sclerosis patients: a population-based study. J Neurol Sci. 2006 Dec 1;250(1-2):45-9. doi: 10.1016/j.jns.2006.06.027. Epub 2006 Aug 22. PMID 16920152
- [Background] Miles A, Huckabee ML. Intra- and inter-rater reliability for judgement of cough following citric acid inhalation. Int J Speech Lang Pathol. 2013 Apr;15(2):209-15. doi: 10.3109/17549507.2012.692812. Epub 2012 Aug 8. PMID 22873621